CLINICAL TRIAL: NCT03188523
Title: A Single-Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Anti-Retroviral Activity of MK-8504 Monotherapy in Anti-Retroviral Therapy (ART)-Naïve, HIV-1 Infected Patients
Brief Title: Activity of MK-8504 in Anti-retroviral-naïve, Human Immunodeficiency Virus 1 (HIV-1) Infected Participants (MK-8504-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8504-002; 2017-000998-37 (EudraCT Number); MK-8504-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-06-14; First posted 2017-06-15 (Actual); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MK-8504 100 mg (Panel A) (Experimental): Participants receive a single oral dose of MK-8504 100 mg.
  Interventions: Drug: MK-8504
- MK-8504 240 mg (Panel B) (Experimental): Participants receive a single oral dose of MK-8504 240 mg.
  Interventions: Drug: MK-8504
- MK-8504 ≤240 mg (Panel C) (Experimental): Participants receive a single oral dose of MK-8504 ≤240 mg.
  Interventions: Drug: MK-8504
- MK-8504 ≤240 mg (Panel D) (Experimental): Participants receive a single oral dose of MK-8504 ≤240 mg.
  Interventions: Drug: MK-8504

INTERVENTIONS:
Drug: MK-8504 — After at least an 8-hour fast, a single oral dose of MK-8504 will be administered in capsule form.

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetics (PK), and anti-retroviral therapy (ART) activity of monotherapy with MK-8504 (a tenofovir pro-drug), in ART-naïve Human Immunodeficiency Virus (HIV)-1 infected participants. The primary hypothesis is that MK-8504, at a dose that is sufficiently safe and well tolerated, has superior antiretroviral activity compared to placebo, as measured by change from baseline in plasma HIV-1 ribonucleic acid (RNA) at 168 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-breast feeding female
* Have a Body Mass Index (BMI) ≤35 kg/m^2
* Other than HIV infection, have stable baseline health based on medical history, physical examination, vital sign measurements, and laboratory safety test
* Is documented HIV-1 positive
* Is diagnosed with HIV-1 infection 3 months prior to screening
* Is ART-naïve
* Has not received an investigational agent or marketed ART within 30 days of study drug administration and is willing to receive no other ART for the duration of this study
* Agree to follow smoking and other trial restrictions

Exclusion Criteria:

* Is mentally or legally institutionalized / incapacitated, has significant emotional problems at the time of pretrial (screening) visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder of the last 5 years
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer (malignancy)
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food
* Is positive for hepatitis B surface antigen
* Has a history of chronic Hepatitis C
* Has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit.
* Has participated in another investigational trial within 4 weeks or 5 half-lives, whichever is greater, prior to the Day 1 Dosing visit
* Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of trial drug, throughout the trial, until the post-trial visit
* Consumes greater than 3 glasses of alcoholic beverages or distilled spirits per day
* Consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day
* Is an excessive smoker (i.e., more than 10 cigarettes/day) and is unwilling to restrict smoking to ≤10 cigarettes per day
* Have clinically significant abnormality on the electrocardiogram (ECG) performed at the prestudy (screening) visit and/or prior to administration of the initial dose of study drug
* Has a positive urine drug screen (except for cannabis) at screening and/or predose, rechecks are allowed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Charite Research Organisation GmbH. ( Site 0002), Berlin, Germany
- St Stephen's Clinical Research ( Site 0001), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve participants infected with Human Immunodeficiency Virus 1 (HIV-1) were enrolled into Panels A and B. Due to an earlier than anticipated achievement of the study primary study objectives, Panels C and D were not conducted and no participants were enrolled in these panels.
Groups:
- MK-8504 ≤240 mg (Panel C); MK-8504 ≤240 mg (Panel D): Participants were to receive a single oral dose of MK-8504 ≤240 mg. This panel did not enroll any participants.
Period: Overall Study
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B) | MK-8504 ≤240 mg (Panel C) | MK-8504 ≤240 mg (Panel D)
Started | 6 | 6 | 0 | 0
Completed | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (6.0) | 35.5 (7.0) | 33.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Baseline Plasma HIV-1 Ribonucleic Acid (RNA) [Mean (Standard Deviation); unit: Log10 copies/mL] | 4.31 (0.34) | 4.60 (0.64) | 4.45 (0.51)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma HIV-1 Ribonucleic Acid (RNA) at 168 Hours Post-Dose
Description: Plasma samples were collected from participants after a single dose of MK-8504 to assess viral load. The log10 plasma HIV-RNA (copies/mL) measurements from participants in each panel were pooled and analyzed based on a longitudinal data analysis model. Change from baseline to 168 hours post-dose was determined for each treatment group. Results are expressed as change in HIV RNA log10 (copies/mL).
Time Frame: Baseline, 168 hours post-dose
Population: All randomized participants
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 (copies/mL)
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
log10 (copies/mL) | -1.06 [-1.49 to -0.62] | -0.95 [-1.38 to -0.51]
Statistical Analysis 1: Comparison: MK-8504 100 mg (Panel A); Adjusted by Placebo data pooled from historical placebo data from recent monotherapy studies in HIV-1 infected participants (NCT00100048, NCT01466985, NCT01152255, and NCT01353898) and fitted with a longitudinal data analysis (LDA) model containing fixed effects for study and time, and a random effect for participants. LS mean (95% confidence interval) for change from baseline at 168 hours post dose of pooled historical placebo was -0.03 log10 copies/mL (-0.14, 0.09); Test type: Superiority; Posterior Mean Difference = -1.03 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8504 and placebo at least 0.5 log10 copies/mL was >98%
Statistical Analysis 2: Comparison: MK-8504 240 mg (Panel B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Posterior Mean Difference = -0.92 — Posterior Probability (PP) of true mean difference in the plasma HIV-1 RNA change from baseline between MK-8504 and placebo at least 0.5 log10 copies/mL was >95%

2. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the Sponsor's product, was also an AE. The number of participants experiencing at least one AE was reported for each arm.
Time Frame: From Day 1 through Post-Trial Visit (up to 25 days)
Population: All participants that received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
Participants | 5 | 6

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the Sponsor's product, was also an AE. The number of participants that discontinued study treatment due to an AE was reported for each arm.
Time Frame: Day 1
Population: All participants that received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

4. Secondary Outcome: Area Under the Concentration-Time Curve of MK-8504 in Plasma From Time 0 to Last Measurable Concentration (AUC0-last)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine AUC0-last of plasma MK-8504. AUC0-last was defined as the area under the concentration time curve of plasma MK-8504 from time 0 to last measurement, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with the study procedure, and had available plasma pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 2.58 (63.4) | 6.20 (32.1)

5. Secondary Outcome: Area Under the Concentration-Time Curve of MK-8504 in Plasma From Time 0 to Infinity (AUC0-inf)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine AUC0-inf of plasma MK-8504. AUC0-inf was defined as the area under the concentration time curve of plasma MK-8504 from time 0 to infinite time, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with the study procedure, and had available plasma PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 2.59 (63.0) | 6.25 (32.0)

6. Secondary Outcome: Area Under the Concentration-Time Curve of MK-8504 in Plasma From Time 0 to 168 Hours (AUC0-168hr)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine AUC0-168hr of plasma MK-8504. Because plasma MK-8504 was expected to rapidly disappear from plasma based on prior experience with healthy participants, sampling was done until 72 hrs and AUC0-168 hr was computed from these data assuming 1) a mono-exponential concentration decline after 72hrs; 2) accurate estimation of the elimination rate based on available data; and 3) no involvement of other processes besides elimination after 72 hrs.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 2.61 (62.4) | 6.26 (32.5)

7. Secondary Outcome: Time to Maximum Concentration of MK-8504 in Plasma (Tmax)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine Tmax of plasma MK-8504. Tmax was defined as the time at which maximum concentration of MK-8504 in plasma was observed, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Full Range); unit: Hour (hr)
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
Hour (hr) | 1.00 [0.50 to 2.00] | 0.75 [0.50 to 1.00]

8. Secondary Outcome: Maximum Concentration of MK-8504 in Plasma (Cmax)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine Cmax of plasma MK-8504. Cmax was defined as the maximum concentration of MK-8504 in plasma observed, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM | 2.72 (81.6) | 5.32 (22.5)

9. Secondary Outcome: Apparent Terminal Half Life of MK-8504 in Plasma (t½)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine t½ of plasma MK-8504. t½ was defined as the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
hr | 3.02 (38.6) | 6.27 (29.7)

10. Secondary Outcome: Apparent Total Clearance of MK-8504 in Plasma (CL/F)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine CL/F of plasma MK-8504. CL/F was defined as the apparent total clearance of the drug from plasma after oral administration, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)/hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
liters (L)/hr | 67.7 (63.0) | 67.4 (32.0)

11. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-8504 in Plasma
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine Vz/F of plasma MK-8504. Vz/F was defined as the apparent volume of distribution of the drug in plasma during the terminal phase after non-intravenous administration, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
liters (L) | 295 (55.1) | 609 (17.8)

12. Secondary Outcome: Intracellular Area Under the Concentration-Time Curve of Tenofovir-Diphosphate (TFV-DP) From Time 0 to 168 Hours (Intracellular AUC0-168hr) In Peripheral Blood Mononuclear Cells (PBMCs)
Description: Blood samples were collected in a fasted state pre- and post-dose, processed for PBMC samples, and used to determine the intracellular AUC0-168hr of TFP-DP in PBMCs. TFV-DP is formed via metabolism of MK-8504 in plasma, PBMC and in other tissues. Intracellular AUC0-168hr was defined as the area under the concentration time curve of TFV-DP in PBMCs from time 0 to 168 hours, following a single dose of MK-8504.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, and 168 hours post-dose
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment, were compliant with the study procedure, and had available PBMC PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 346 (22.5) | 885 (17.8)

13. Secondary Outcome: Intracellular Area Under the Concentration-Time Curve of Tenofovir-Diphosphate (TFV-DP) From Time 0 to Infinity (Intracellular AUC0-inf) In Peripheral Blood Mononuclear Cells (PBMCs)
Description: Blood samples were collected in a fasted state pre- and post-dose, processed for PBMC samples, and used to determine the intracellular AUC0-inf of TFV-DP in PBMCs. TFV-DP is formed via metabolism of MK-8504 in plasma, PBMC and in other tissues. Intracellular AUC0-inf was defined as the area under the concentration time curve of TFV-DP in PBMCs from time 0 to infinite time, following a single dose of MK-8504.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, 168, 240, 384, and 600 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 433 (22.9) | 1020 (19.3)

14. Secondary Outcome: Intracellular Time to Maximum Concentration (Intracellular Tmax) of Tenofovir-Diphosphate (TFV-DP) In Peripheral Blood Mononuclear Cells (PBMCs)
Description: Blood samples were collected in a fasted state pre- and post-dose, processed for PBMC samples, and used to determine the intracellular Tmax of TFV-DP. TFV-DP is formed via metabolism of MK-8504 in plasma, PBMC and in other tissues. Intracellular Tmax was defined as the time at which maximum intracellular concentration of TFV-DP in PBMCs was observed, following a single dose of MK-8504.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, 168, 240, 384, and 600 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Full Range); unit: hours (hr)
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
hours (hr) | 4.00 [4.00 to 12.00] | 12.00 [4.00 to 24.00]

15. Secondary Outcome: Intracellular Maximum Concentration (Intracellular Cmax) of Tenofovir-Diphosphate (TFV-DP) In Peripheral Blood Mononuclear Cells (PBMCs)
Description: Blood samples were collected in a fasted state pre- and post-dose, processed for PBMC samples, and used to determine the intracellular Cmax of TFV-DP. TFV-DP is formed via metabolism of MK-8504 in plasma, PBMC and in other tissues. Intracellular Cmax was defined as the maximum intracellular concentration of TFV-DP in PBMCs observed, following a single dose of MK-8504.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, 168, 240, 384, and 600 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM | 5.89 (22.3) | 15.1 (52.6)

16. Secondary Outcome: Intracellular Apparent Terminal Half Life (Intracellular t½) of Tenofovir-Diphosphate (TFV-DP) In Peripheral Blood Mononuclear Cells (PBMCs)
Description: Blood samples were collected in a fasted state pre- and post-dose, processed for PBMC samples, and used to determine the intracellular t½ of TFV-DP. TFV-DP is formed via metabolism of MK-8504 in plasma, PBMC and in other tissues. Intracellular t½ was defined as the time required to divide the intracellular concentration by two after reaching pseudo-equilibrium, following a single dose of MK-8504.
Time Frame: Pre-dose, 4, 12, 24, 48, 72, 96, 168, 240, 384, and 600 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
hour (hr) | 72.4 (21.5) | 67.5 (42.1)

17. Secondary Outcome: Intracellular Concentration of Tenofovir-Diphosphate (TFV-DP) at 168 Hours (Intracellular C168hr) In Peripheral Blood Mononuclear Cells (PBMCs)
Description: Blood samples were collected in a fasted state, processed for PBMC samples, and used to determine the intracellular C168hr of TFV-DP. TFV-DP is formed via metabolism of MK-8504 in plasma, PBMC and in other tissues. Intracellular C168hr was defined as the intracellular concentration of TFV-DP in PBMCs at 168 hours, following a single dose of MK-8504.
Time Frame: 168 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM | 0.910 (19.4) | 1.35 (24.7)
Statistical Analysis 1: Comparison: MK-8504 100 mg (Panel A); PBMC TFV-DP C168hr values pooled, natural log transformed and analyzed based on a linear model containing a fixed effect for dose level. The posterior probability that the true GM of PBMC TFV-DP C168hr level was ≥0.1 μM was calculated for the dose level using flat priors under a normal likelihood assumption. An 80% posterior probability for a dose level that also exhibits acceptable safety and tolerability would satisfy the secondary PK hypothesis; Test type: Other; Posterior Probability (percentage) = 99 — Posterior Probability (percentage) of true geometric mean (GM) C168hr TFV-DP level in PBMCs ≥0.1 μM
Statistical Analysis 2: Comparison: MK-8504 240 mg (Panel B); [analysis description as in outcome 17, analysis 1]; Test type: Other; Posterior Probability (percentage) = 99 — Posterior Probability (percentage) of true geometric mean (GM) C168hr TFV-DP level in PBMCs ≥0.1 μM

18. Secondary Outcome: Area Under the Concentration-Time Curve of Tenofovir in Plasma From Time 0 to Last Measurable Concentration (AUC0-last)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine AUC0-last of plasma tenofovir. AUC0-last was defined as the area under the concentration time curve of plasma tenofovir from time 0 to last measurement, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 1.71 (19.5) | 4.47 (14.2)

19. Secondary Outcome: Area Under the Concentration-Time Curve of Tenofovir in Plasma From Time 0 to Infinity (AUC0-inf)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine AUC0-inf of plasma tenofovir. AUC0-inf was defined as the area under the concentration time curve of plasma tenofovir from time 0 to infinite time, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 2.19 (27.6) | 6.00 (19.6)

20. Secondary Outcome: Area Under the Concentration-Time Curve of Tenofovir in Plasma From Time 0 to 168 Hours (AUC0-168hr)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine AUC0-168hr of plasma tenofovir. Because plasma tenofovir was expected to rapidly disappear from plasma based on prior experience with healthy participants, sampling was done until 72 hrs and AUC0-168 hr was computed from these data assuming 1) a mono-exponential concentration decline after 72hrs; 2) accurate estimation of the elimination rate based on available data; and 3) no involvement of other processes besides elimination after 72 hrs.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM·hr | 2.13 (25.7) | 5.72 (17.3)

21. Secondary Outcome: Time to Maximum Concentration of Tenofovir in Plasma (Tmax)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine Tmax of plasma tenofovir. Tmax was defined as the time at which maximum concentration of tenofovir in plasma was observed, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Full Range); unit: Hour (hr)
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
Hour (hr) | 2.00 [1.00 to 2.00] | 2.00 [2.00 to 2.00]

22. Secondary Outcome: Maximum Concentration of Tenofovir in Plasma (Cmax)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine Cmax of plasma tenofovir. Cmax was defined as the maximum concentration of tenofovir in plasma observed, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
μM | 0.0727 (25) | 0.156 (22.8)

23. Secondary Outcome: Apparent Terminal Half Life of Tenofovir in Plasma (t½)
Description: Plasma samples were collected in a fasted state pre- and post-dose and used to determine t½ of plasma tenofovir. t½ was defined as the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, following a single dose of MK-8504.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 12, 24, 36, 48, and 72 hours post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
Number analyzed (Participants) | 6 | 6
hr | 32.3 (23.7) | 35.3 (29.0)

ADVERSE EVENTS:
Time Frame: From Day 1 through Post-Trial Visit (up to 25 days)
Description: All participants that received at least one dose of treatment.
Arm/Group | MK-8504 100 mg (Panel A) | MK-8504 240 mg (Panel B)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8504 100 mg (Panel A) (N=6) | MK-8504 240 mg (Panel B) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 3 (6)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT03188523/Prot_SAP_000.pdf